CLINICAL TRIAL: NCT04946331
Title: Comparison of Lung Function Based on Electrical Impedance Tomography and CT Lung Volume in Patients With Rib Fractures
Acronym: EIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 202103085RIPC
Record Dates: First submitted 2021-06-23; First posted 2021-06-30 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-06

CONDITIONS: Rib Fractures
Keywords: Pulmonary function; Electrical impedance tomography system
MeSH Terms: conditions — Rib Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): participants receive no surgical treatment
  Interventions: Device: Electrical impedance tomography system
- Rib Fixation Surgery (Experimental): participants receive surgical treatment
  Interventions: Device: Electrical impedance tomography system

INTERVENTIONS:
Device: Electrical impedance tomography system — Which can use the applied current and measurement voltage through the body surface electrode group, and use the reconstruction algorithm to construct an image imaging system that exceeds the cross-sectional, which can provide images of the internal physiological changes of the chest contour, in order to quantify the changes in lung function caused by rib fractures.
  Other Names: EIT

SUMMARY:
Our research uses the electrical impedance tomography system (EIT), which can use the applied current and measurement voltage through the body surface electrode group, and use the reconstruction algorithm to construct an image imaging system that exceeds the cross-sectional, which can provide images of the internal physiological changes of the chest contour, in order to quantify the changes in lung function caused by rib fractures.

DETAILED DESCRIPTION:
Rib fractures are one of the most common injuries following blunt trauma, occurring in approximately 10% of all trauma patients. Rib fracture injuries extend across a broad spectrum of severity from a single fractured rib which may be sustained in a fall or sporting injury, to multiple fractured ribs resulting in a flail chest with paradoxical chest wall movement and respiratory failure.

Flail chest, which defines multiple adjacent ribs broken in multiple places, is the most serious chest injury, and it damages the chest wall integrity and causes "paradoxical motion" from the detachment of a segment from the rest of the chest wall. Surgical management of rib fractures has received increasing attention in recent years with the development of new fixation techniques.

The mortality rate is 4% to 20%. Flail chest (FC), which defines multiple adjacent ribs broken in multiple places, is the most serious chest injury, and it damages the chest wall integrity and causes "paradoxical motion" from the detachment of a segment from the rest of the chest wall. Pulmonary contusion (PC) is the most common chest injury. These conditions frequently exist at the same time. Currently, a deeper understanding of FC pathophysiology exists, and its management has evolved substantially over the past 6 decades.

The earliest treatment for FC was surgery. With the increasing technological advancements available in the intensive care unit, conservative management, based on mechanical ventilation supplemented with intensive pain control, has become more common. Using positive airway pressure to reduce the asynchronous movement of FC could avoid surgical risks and postoperative complications. Conservative treatment has been administered frequently in previous years.

A growing number of researchers have found that surgery for FC could reduce the duration of mechanical ventilation, the ICU length of stay, the hospital length of stay, the incidence of pneumonia and tracheostomy, and mortality. Additional benefits included decreased doses of analgesic and sedative drugs and avoidance of thoracic deformity, and patients could return to previous employment quicker than could those treated conservatively.

Therefore, the improvement of lung function is a key indicator for the treatment of rib fractures and thoracic trauma, because lung function is related to lung expansion, chest wall stability, and thoracic deformation, which can lead to pneumonia, respiratory failure, difficult weaning, and prolong hospitalization. However, traditional pulmonary function measurement is based on an Incentive Spirometry. This examination requires the cooperation of the patient and also requires sufficient space and equipment. It is not suitable for acute trauma patients in intensive care units. In addition, the induced spirometer can only measure respiratory parameters such as vital capacity. It cannot locate and monitor the collapse part of lung and the range of pulmonary atelectasis. It must rely heavily on computer tomography and other imaging assistance, which is very unsatisfactory. Therefore, how to simultaneously develop an effective monitoring method for lung function and lung expansion is the current top priority.

For these reason, our research uses the electrical impedance tomography system (EIT), which can use the applied current and measurement voltage through the body surface electrode group, and use the reconstruction algorithm to construct an image imaging system that exceeds the cross-sectional, which can provide images of the internal physiological changes of the chest contour, in order to quantify the changes in lung function caused by rib fractures.

This study is a combine research project of patients from the Department of Traumatology of National Taiwan University Hospital and the Department of Traumatology of Far Eastern Memorial Hospital. The study is expected to be collected from July 2021 to December 2022 for one and a half years. Hospitalized patients with traumatic rib fractures were collected and analyzed in a prospective study method, and the patients with internal rib fractures in Far Eastern Memorial Hospital were collected and analyzed, and their lung function changes after the operation will be tracked.

ELIGIBILITY:
Inclusion Criteria:

1. Over 20 years old
2. At least 3 rib fractures due to thoracic trauma, or in compliance with the definition of flail chest.
3. Consciousness Coma Index (GSC) 14 points or above

Exclusion Criteria:

1. Consciousness coma index (GSC) less than 14 points
2. BMI> 50
3. Have received thoracic surgery (including patients with partial and full lobes)
4. Patients with pacemakers
5. Spinal lesions or fractures of spinal instability
6. Vulnerable population
7. Patients who need to remove more than one lung lobe during surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
1st EIT test | In 72 hours
  Pulmonary function test with EIT before surgical in 72 hrs
2nd EIT test | In 2nd weeks
  Pulmonary function test with EIT after surgical / (no surgical ) in 2nd weeks
3rd EIT test | In 12th weeks
  Pulmonary function test with EIT after surgical / (no surgical ) in 12th weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Chi Liao, MD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan